CLINICAL TRIAL: NCT07359521
Title: Implementation and Evaluation of a Complex Intervention to Reduce Avoidable Transitions Between Nursing Home and Hospital (RATHER-NH): Study Protocol for a Pilot Cluster Randomized Controlled Trial.
Brief Title: Implementation and Evaluation of a Complex Intervention to Reduce Avoidable Transitions Between Nursing Home and Hospital
Acronym: RATHER-NH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25441_RATHER-NH RCT; G069022N (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2025-12-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Potentially Avoidable Hospitalisations
Keywords: Nursing homes; Potentially avoidable hospitalisations; Quality improvement program; Implementation; Pilot cluster RCT

STUDY DESIGN:
Intervention Model Description: Pilot Cluster RCT with an embedded process evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Nursing homes in the intervention group will implement tools from the RATHER-NH intervention toolkit using a tailored implementation strategy over a period of approximately 9 months.
  Interventions: Other: RATHER-NH Toolkit
- Control group (No Intervention): Care as usual

INTERVENTIONS:
Other: RATHER-NH Toolkit — 1. Quality Improvement Tool for Review of Acute Care Transfers
  2. Stop and Watch Early Warning Tool
  3. SBAR Communication Form
  4. Engaging Your Hospitals - Tip Sheets
  5. Care paths
  6. Advance care planning document
  7. 'In the moment' communication tool
  Arms: Intervention group

SUMMARY:
Hospital admissions can have a negative impact on the physical and emotional health of nursing home residents. Although evidence-based interventions have been developed to reduce hospitalisations, the evidence regarding their effectiveness is inconclusive and challenges have been reported in implementing these interventions within the nursing home context. Hence, this study aimed to implement and evaluate a complex intervention to reduce avoidable transitions between nursing home and hospital (RATHER-NH).

DETAILED DESCRIPTION:
The researchers will conduct a pilot cluster randomized controlled trial (RCT) of the RATHER-NH intervention with an embedded process evaluation. This study has two specific objectives: 1) to evaluate the implementation of the RATHER-NH intervention, the perceived impact and underlying mechanisms of impact, and the contextual factors influencing implementation and impact; and 2) To assess the feasibility of the trial methods and procedures, and the potential primary and secondary outcome measures for a future full-scale RCT.

The study will be conducted in twelve nursing homes in Flanders, of which six will be randomly assigned to the intervention group and six to the control group.

The researchers will use the MRC guidance on complex intervention development and evaluation combined with the integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) framework to guide the implementation and evaluation of RATHER-NH.

Based on the results of the qualitative study with nursing home residents, family carers and professional stakeholders, and on existing scientific literature, a first version of a logic model was developed, which illustrates the different determinants and mechanisms that influence the anticipated outcomes and impact of the RATHER-NH intervention. The logic model was used to select relevant intervention tools from the INTERACT Quality Improvement Program, the VZP+ project and our own self-developed tool concerning 'in the moment' communication tool:

A) Quality Improvement Tool for Review of Acute Care Transfers This tool can help nursing home staff members to reflect on the decision-making process to hospitalise a nursing home resident.

B) Stop and Watch Early Warning Tool This is a checklist that marks the most relevant changes in the physical and behavioural condition of a nursing home resident that eventually may lead to a potentially avoidable hospitalisation.

C) SBAR Communication Form The SBAR Communication Form ("Situation - Background - Assessment - Recommendation") is a tool designed to help nursing home staff efficiently brief their colleagues about a resident's condition at the start of a shift.

D) Engaging Your Hospitals - Tip Sheets This is a list with tips and tricks for nursing homes to improve communication with nearby hospitals.

E) Care paths Care paths have been developed for several Ambulatory Care Sensitive Conditions (ACSCs), which are conditions that can lead to unplanned hospitalisation which may be avoided if the condition is promptly detected and managed correctly through access to medical care in the nursing home.

F) Advance care planning document The advance care planning (ACP) document has been selected from the VZP+ project, which aims to support nursing home staff in conducting and documenting advance care planning discussions with residents and their family carers.

G) 'In the moment' communication tool This tool does not only cover communication with the general practitioner but also with the resident, family members and other nursing home staff members.

The tools from the RATHER-NH intervention toolkit have fixed and flexible elements. To adapt elements of the tools to the local context, each participating nursing home will engage in a facilitated group discussion to assess the context and their specific needs, facilitated by the researcher and guided by the i-PARIHS framework. While the fixed elements of each tool need to be maintained to preserve the intervention fidelity, the flexible and hence adaptable elements can be tailored to fit the specific needs, routines, and structures of each nursing home. This ensures that the intervention is both evidence-informed and context-sensitive, increasing the likelihood of successful implementation.

Based on evidence from our qualitative study with key stakeholders and findings from other relevant studies, several implementation barriers are anticipated when implementing complex nursing home interventions such as the RATHER-NH intervention. These barriers were linked to the implementation strategies as described in the Expert Recommendations for Implementing Change (ERIC) Matching Tool. These strategies combined will form the implementation strategy for RATHER-NH (e.g. conduct educational meetings, ongoing training and identify and prepare champions). To ensure the implementation strategy is responsive to the specific needs of each nursing home, this will also be discussed during the facilitated group discussion to tailor and operationalise the implementation strategies by adapting the flexible elements of the implementation strategies to the local context. Next to the researcher, an external trainer will be recruited to support the implementation of the intervention within the nursing homes.

ELIGIBILITY:
Inclusion criteria for nursing homes:

* A capacity of at least 60 beds
* Active engagement for the study from nursing home management, head nurses and the coordinating & advisory physician, meaning:

  1. The nursing home manager, head nurses and the coordinating & advisory physician agree that the implementation of the RATHER-NH intervention is a priority for their facility.
  2. The nursing home manager agrees to provide time for the nursing home staff members to participate in activities related to the implementation of RATHER-NH such as attending information sessions, training workshops, and feedback moments.
  3. The nursing home manager is willing to allocate time to at least two nursing home staff members (each approximately 0.1 FTE for the study duration) to act as local project champions and to at least four other staff members (type of staff to be decided with the nursing home manager) to form a local action team to support the implementation and evaluation of RATHER-NH.

Exclusion criteria for nursing homes:

* Already participated in another project designed to reduce potentially avoidable hospitalisations.
* Already taking part in another major quality improvement initiative or study.
* A large reorganisation or change in staff is taking place or is planned during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Outcomes on healthcare use per 100 person-months | Retrospective baseline measurement of 3 months, during the intervention (period of 9 months) untill 3 months post-intervention for the post-interventions measurement.
  Rate of hospitalisations per 100 person-months, rate of out-of-hours GP contacts per 100 person-months, rate of emergency department visits (without hospitalisation) per 100 person-months.
Outcomes on healthcare use per hospitalisation | Retrospective baseline measurement of 3 months, during the intervention (period of 9 months) untill 3 months post-intervention for the post-interventions measurement.
  Length of hospital stay, cause of hospitalisation, hospitalisation in the last month of life (in case of death) and place of death

SECONDARY OUTCOMES:
Self-Efficacy and Outcome Expectancy Scales for Job-Related applications questionnaire to measure the job-related self-efficacy of nursing home staff members on a 7-point Likert Scale | During the retrospective baseline measurement of 3 months and during the 3 months post-intervention measurement.
  Staff self-efficacy will be measured through the validated 31-item Self-Efficacy and Outcome Expectancy Scales for Job-Related applications questionnaire, which involves four sub-scales (i.e. personal efficacy beliefs scale, personal outcome expectancy scale, collective efficacy beliefs scale, collective outcome expectancy scale) on a 7-point Likert Scale.

OTHER OUTCOMES:
Process outcome: Notes of facilitated group discussions on implementation strategies using a framework analysis | During the pre-implementation phase of the intervention (first 3 months of the 9 month intervention period)
  The researcher will take notes during the facilitated group discussions in which the implementation strategies are adapted and tailored according to the specific needs and context of the nursing homes. A framework analysis will be used to analyse the data.
Process outcome: Case studies to examine the perspectives on the decision-making process prior to an unplanned hospitalisation using a cross-case analysis | During the intervention (period of 9 months)
  Multiple case studies will be conducted using semi-structured interviews to examine the decision-making process prior to an unplanned hospitalisation.
  In every participating nursing home, 2 case studies will be conducted.
  For every case, semi-structured interviews will be conducted with:
  1. the nurse most involved in the hospitalisation decision
  2. the resident's GP or other physician involved in the hospitalisation decision
  3. the resident and/or a family member, where feasible. A cross-case analysis will be used to analyse the data.
Process outcome: Minutes of action team meetings on the implementation process using a content analysis | During the intervention (period of 9 months)
  The action teams will be asked, including the local project champions, to take minutes of their meetings to discuss the implementation process. Afterwards, the data of all the participating nursing homes will be compared in order to evaluate whether are not there were major differences between facilities regarding the topics that were discussed or challenges they experienced. A content analysis will be used to analyse the data.
Process outcome: Structured diaries on the use of the intervention tools, pre-implementation and implementation strategies using a content anaysis | During the intervention (period of 9 months)
  To evaluate how the intervention tools were used, and how the pre-implementation and implementation strategies were delivered, the local project champions, trainer and researcher will be asked to keep diaries. Afterwards, the data of all the participating nursing homes will be compared in order to evaluate whether are not there were major differences between facilities regarding the use of the intervention tools and the used pre-implementation and implementation strategies. A content analysis will be used to analyse the data.
Process outcome: Semi-structured focus groups on the relevance, acceptability and feasibility of the intervention tools and the used implementation strategies using a framework analysis | During the 3 months post-intervention measurement
  1. Semi-structured focus group with the action team members to explore their experiences with the RATHER-NH intervention tools, pre-implementation strategies and implementation strategies.
  2. Semi-structured focus group with a selection of nursing staff who were not part of the action team to explore their experiences with the RATHER-NH intervention tools, pre-implementation strategies and implementation strategies. Next to this, it will be evaluated to which extent the intervention was known by nursing home staff members that were not active members of the study.
  3. Semi-structured interviews with the local project champions to explore their experiences with the RATHER-NH intervention tools, pre-implementation strategies and implementation strategies.
  A framework analysis will be used to analyse the data.
Process outcome: Perceived impact of the intervention and the underlying mechanisms of impact using the 'most significant change' technique | During the 3 months post-intervention measurement
  Nursing home staff members will be invited to provide short written stories about the most significant change that they experienced related to the intervention, why this was the most significant change according to them and how and why these changes happened according to them. The stories will be collected and discussed among the action team members and local champions during one of the action team meetings. Through this in-depth group discussion, the most significant stories will be selected, including documentation of reasons why these were considered as most significant according to the group.
Feasibility outcome: Self-structured study logs kept by researcher using a content analysis | During the intervention (period of 9 months)
  The researcher will continuously document information on the recruitment, retention, data collection methods and trial procedures in a self-structured study log during the study. This log book will be used to evaluate the used strategies and procedures in order to decide whether or not these are useful in a future full-scale RCT. A content analysis will be used to analyse the data.
Feasibility outcome: Semi-structured interviews on the acceptability of the recruitment strategies, randomisation procedures and data collection processes using a framework analysis | During the 3 months post-intervention measurement
  Semi-structured interviews will be conducted with the managers and key contact persons of the participating nursing homes to explore their perception on the acceptability of the recruitment procedures, the study retention, the randomisation process, the data collection processes and the challenges related to the trial methods. A framework analysis will be used to analyse the data.
Review of returned questionnaires and registration documents on their completeness | During the 3 months post-intervention measurement
  The researcher will review the returned self-efficacy questionnaires and healthcare use registration documents regarding their completeness. More specifically, the researcher will assess the number and type of missing/incomplete responses in each of the questionnaires and registration forms. This will be used to evaluate whether the used strategies to promote staff members to fill in the questionnaire is feasible in a future full-scale RCT.

CONTACTS AND LOCATIONS:
Overall Officials: Tinne Smets, Prof., Principal Investigator — End-of-Life Care Research Group - Vrije Universiteit Brussel en Universiteit Gent

IPD SHARING:
Plan to Share IPD: No
IPD will not be collected during the trial. The collected data will be on facility level.